CLINICAL TRIAL: NCT02653599
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Parallel-Group Multi-Center Study to Evaluate the Efficacy and Safety of TTP273 Following 12 Weeks Administration in Subjects With Type 2 Diabetes Mellitus on a Stable Dose of Metformin
Brief Title: A Study to Evaluate Safety and Efficacy of TTP273 for 12 Weeks in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTP273-201
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TTP273 300 mg daily (150 mg BID) (Experimental): Two 75 mg tablets of TTP273 administered orally twice daily for 12 weeks
  Interventions: Drug: TTP273
- TTP273 150 mg daily (Experimental): Two 75mg tablets of TTP273 administered orally once daily and two placebo tablets administered orally once daily for 12 weeks
  Interventions: Drug: TTP273; Drug: Placebo
- Placebo (Placebo Comparator): Two matching placebo tablets administered orally twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTP273
  Arms: TTP273 150 mg daily; TTP273 300 mg daily (150 mg BID)
Drug: Placebo
  Arms: Placebo; TTP273 150 mg daily

SUMMARY:
This trial is a multi-center, randomized, double-blind, placebo-controlled parallel group, Phase 2 study in subjects with Type 2 diabetes mellitus on a stable dose of metformin to evaluate the safety and efficacy of TTP273 versus placebo glucose control and body weight following administration for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a 6 month diagnosis of Type 2 diabetes mellitus prior to screening and meets the American Diabetes Association (ADA) guidelines for Type 2 diabetes mellitus.
* On a stable regimen of metformin monotherapy equivalent to at least 1000 mg/day for the last 3 months prior to screening.
* Males. Females of non-childbearing potential.
* Generally stable health without a history of major surgery or significant injuries within the last year and without an active infection.

Exclusion Criteria:

* Diagnosis of Type 1 diabetes mellitus, maturity-onset diabetes of the young, insulin-requiring Type 2 Diabetes, other unusual or rare forms of diabetes mellitus, or history of diabetic ketoacidosis.
* Participation in a clinical trial and receipt of an investigational product within 30 days.
* Participation in any formal weight loss program, or fluctuation of > 5% in body weight, or having received medications approved for weight loss within 3 months prior to screening or contemplating such therapy during the trial.
* Previous surgical treatment of obesity.
* Have a history of hypoglycemic episode requiring glucose, glucagon, or orange juice administered by someone other than the patient within 6 months prior to screening.
* Use of other diabetic agents except metformin within 3 months prior to Screening.
* History of pancreatitis.
* Blood donation of approximately 1 pint (500 mL) within 8 weeks prior to screening.
* History of hemolytic anemia, chronic transfusion requirement or other condition rendering HbA1c results unreliable.
* History of MEN-2 or family history of medullary thyroid cancer.
* History or presence of clinically significant disease (other than Type 2 diabetes mellitus).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline at 12 weeks | Day 1 to Week 12

SECONDARY OUTCOMES:
Percentage of subjects who achieve HbA1c <7% at 12 weeks | Day 1 to Week 12
Change in body weight from baseline at 12 weeks | Day 1 to Week 12
Change in plasma glucose levels from baseline at 12 weeks | Day 1 to Week 12
Change in lipid Levels from baseline at 12 weeks | Day 1 to Week 12
Change in insulin levels from baseline at 12 weeks | Day 1 to Week 12
Change in C-peptide levels from baseline at 12 weeks | Day 1 to Week 12
Adverse Events | Day 1 to Week 14
Blood Pressure | Day 1 to Week 14
Electrocardiogram Parameters | Day 1 to Week 14
Hematology | Day 1 to Week 14
Blood Chemistry | Day 1 to Week 14
Urinalysis | Day 1 to Week 14
Pulse | Day 1 to Week 14

OTHER OUTCOMES:
Change in glucagon levels from baseline at 12 weeks | Day 1 to Week 12
Change in glucagon-like peptide-1 levels from baseline at 12 weeks | Day 1 to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Freeman, Ph.D., Study Chair — vTv Therapeutics LLC
Locations (28):
- United States (28):
  - Costa Mesa, California
  - Encino, California
  - Huntington Park, California
  - Los Angeles, California
  - Oakland, California
  - Sacramento, California
  - DeLand, Florida
  - Miami Lakes, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Evanston, Illinois
  - Flint, Michigan
  - Omaha, Nebraska
  - The Bronx, New York
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Morehead City, North Carolina
  - Cincinnati, Ohio
  - Norman, Oklahoma
  - Corpus Christi, Texas
  - Houston, Texas
  - Humble, Texas
  - Hurst, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Richland, Washington